CLINICAL TRIAL: NCT02789254
Title: First in Man Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of the Fc-optimized FLT3 Antibody FLYSYN for the Treatment of Acute Myeloid Leukemia Patients With Minimal Residual Disease
Brief Title: FLYSYN in MRD Positive AML
Acronym: FLYSYN-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synimmune GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLYSYN_Version 6.1-17.09.2019
Record Dates: First submitted 2016-05-13; First posted 2016-06-02 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; Fms-like receptor tyrosine kinase (FLT3); stem cell transplantation; complete remission; CD135; antibodies; Leukemia; AML; Fc-optimized
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Pathologic Complete Response; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: FLYSYN (Experimental): IV infusion over a 3-hr duration
  Interventions: Biological: FLYSYN

INTERVENTIONS:
Biological: FLYSYN — Cohort 1:
  Patient 1-3: FLYSYN 0.5 mg/m² BSA* day 1
  Cohort 2:
  Patient 4-6: FLYSYN 0.5 mg/m² BSA day 1 FLYSYN 1.0 mg/m² BSA day 2
  Cohort 3:
  Patient 7-9: FLYSYN 0.5 mg/m² BSA day 1, FLYSYN 4.5 mg/m² BSA day 2
  Cohort 4:
  Patient 10-12 and 13-18: FLYSYN 0.5 mg/m² BSA day 1, FLYSYN 14.5 mg/m² BSA day 2
  Cohort 5:
  Patient 19-21: FLYSYN 0.5 mg/m² BSA day 1, FLYSYN 44.5 mg/m² BSA day 2
  Cohort 6:
  Patient 22-24 and 25-31: FLYSYN 0.5 mg/m² BSA day 1, FLYSYN 14.5 mg/m² BSA day 2, FLYSYN 15 mg/m² BSA day 15, FLYSYN 15 mg/m² BSA day 29
  * The maximum upper limit for calculation of antibody dose is fixed at a body surface of 2.0 m², even if the calculated body surface exceeds this. In this study DLT are defined as the following treatment-related adverse events or laboratory abnormalities, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03.

SUMMARY:
This is a first in human, prospective, multicentric, nonrandomized, open-label study to investigate the safety, tolerability, preliminary efficacy, pharmacokinetics, pharmacodynamics and immunogenicity of the Fc-optimized antibody FLYSYN as monotherapy in adult subjects.

DETAILED DESCRIPTION:
Cohort 1:

Patient 1-3: FLYSYN 0.5 mg/m² body surface area (BSA) day 1

Cohort 2:

Patient 4-6: FLYSYN 0.5 mg/m² body surface area (BSA) day 1 FLYSYN 1.0 mg/m² BSA day 2

Cohort 3:

Patient 7-9: FLYSYN 0.5 mg/m² body surface area (BSA) day 1, FLYSYN 4.5 mg/m² BSA day 2

Cohort 4:

Patient 10-12 and 13-18: FLYSYN 0.5 mg/m² body surface area (BSA) day 1, FLYSYN 14.5 mg/m² BSA day 2

Cohort 5:

Patient 19-21: FLYSYN 0.5 mg/m² body surface area (BSA) day 1, FLYSYN 44.5 mg/m² BSA day 2

Cohort 6:

Patient 22-24 and 25 -31: FLYSYN 0.5 mg/m² body surface area (BSA) day 1, FLYSYN 14.5 mg/m² BSA day 2, FLYSYN 15 mg/m² BSA day 15, FLYSYN 15 mg/m² BSA day 29

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of voluntarily signing an IEC-approved informed consent, there is no upper age limit
* Diagnosis of AML according to WHO criteria
* Confirmed FLT3 expression on leukemic cells
* Known mutational status of FLT3 (FLT3-ITD, FLT3-TKD, FLT3 wild type)
* Hematological CR (ANC count >1.000/μL, Thrombocytes > 100.000/μL), but MRD positivity (determined by NGS and NPM1 RT-PCR, where applicable) after any therapy except allogeneic stem cell transplantation
* Life expectancy of > 3 months
* ECOG performance status ≤ 2
* Subject must be willing to receive transfusion of blood products
* Be willing and able to comply with the study protocol for the duration of the study
* Females of childbearing potential (FCBP) must undergo repetitive pregnancy testing (serum or urine) and results must be negative
* Reliable contraception should be maintained throughout the study and for 6 months after study treatment
* Unless practicing complete abstinence from heterosexual intercourse, sexually active FCBP must agree to use adequate contraceptive methods
* Males (including those who have had a vasectomy) must use an effective barrier method of contraception throughout the study and for 6 months after study treatment if sexually active with a female of childbearing potential
* All subjects must:

  * understand that the investigational product could have a potential teratogenic risk.
  * be counseled about pregnancy precautions and risks of fetal exposure.
  * be able to comply with all study-related procedures, medication use, and evaluations.

Exclusion Criteria:

The presence of ANY of the following criteria will exclude a patient from study enrollment:

* Patients proceeding to hematopoietic stem cell transplantation (suitable candidate and donor available, informed consent of patient)
* Pregnant or breast feeding females
* >5% blasts in bone marrow or extramedullary disease
* Treatment with monoclonal antibody within 3 months before treatment with FLYSYN or known immunoglobulin intolerance
* Known positivity for HIV, active HBV, HCV, or Hepatitis A infection
* No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician and/or other physicians involved in the treatment about study participation
* No consent for biobanking
* Presence of any medical/psychiatric condition or laboratory abnormalities which may limit full compliance with the study, increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Prior history of malignancies, other than AML/MDS, unless the subject has been free of the disease for ≥ 2 years. Exceptions include the following: Basal cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, histological finding of prostate cancer of TNM stage T1
* Patients receiving any medication listed in the Appendix IV "Prohibited Medications" (within 14 days prior to the first dose of study drug)
* Uncontrolled infection, e.g. infection progressing under adequate antimicrobial/antifungal/antiviral treatment
* Patients under ongoing treatment with another investigational medication or having been treated with an investigational medication within 14 days of screening
* Current treatment with immunosuppressive agents
* Systemic diseases (cardiovascular, renal, hepatic, etc.) that would prevent study treatment (e.g., creatinine >1.5x upper normal serum level; bilirubin, AST or AP >2.5x upper normal serum level; heart failure NYHA III/IV; severe obstructive or restrictive ventilation disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE) (CTCAE V 4.03) | until 28 days (i.e. Visit7, day 29) after last dosing

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AE) (CTCAE V 4.03) | until 180 days (i.e.Visit 11, day 180) after last dosing
Pharmacokinetics and pharmacodynamics | Visit 1 to 13
Immunogenicity of FLYSYN based on both absolute (number and percentage of subjects who develop HAMA/HAHA) and semi-quantitative (HAMA/HAHA titer determination of confirmed positive samples) assessments | BSL; Visits 5-7;9-13
Absolute and percent change from baseline in measurements of B, T, and NK cell populations and activation | Visits 1;3;4;5;9
  For evaluation of the status of the immune system, B, T, and NK cells will be measured frequently throughout the study (immune status). The percentage and absolute numbers as well as the absolute and percent changes from baseline of NK cells will be evaluated (determination of absolute NK cell numbers). If feasible, CD16 and CD69 expression on NK cells will be evaluated at baseline and after antibody exposition (NK cell activation). Pending sample availability, endogenous antibody titers (e.g., tetanus titers) will be measured from remaining PK back-up samples in order to gain information about the influence of FLYSYN treatment on normal plasma cells and immunity.
Change in cytokines from baseline | Visits 1-3;5 +6
Overall response rate, defined as MRD negativity or reduction of at least one log step, | BSL; Visits1;4-13
Duration of response, time to MRD progression (log step), time to relapse | BSL; Visits1;4-13
Absolute change from baseline in overall quality of life scores (EORTC QLQ C-30) | Visit 1, Visit 6,Visit 9,Visit 10, Visit 11, Visit 12, Visit 13

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Salih, Prof. Dr., Principal Investigator — Department of Internal Medicine, Internal Medicine II; Oncology, haematology, clinical immunology, rheumatology and pneumology University Hospital Tuebingen
Locations (5):
- Germany (5):
  - University Hospital Tuebingen, Tübingen, Baden-Wurttemberg
  - University Hospital Ulm, Ulm, Baden-Wurttemberg
  - Hannover Medical School, Hanover, Lower Saxony
  - University Hospital of Heidelberg, Heidelberg
  - University of Leipzig Medical Center, Leipzig

IPD SHARING:
Plan to Share IPD: Undecided
publication

REFERENCES:
- [Result] Heitmann JS, Schlenk RF, Dorfel D, Kayser S, Dohner K, Heuser M, Thol F, Kapp-Schwoerer S, Labrenz J, Edelmann D, Marklin M, Vogel W, Bethge W, Walz JS, Grosse-Hovest L, Steiner M, Jung G, Salih HR. Phase I study evaluating the Fc-optimized FLT3 antibody FLYSYN in AML patients with measurable residual disease. J Hematol Oncol. 2023 Aug 17;16(1):96. doi: 10.1186/s13045-023-01490-w. PMID 37587502